CLINICAL TRIAL: NCT07155161
Title: Relationship Backwalking Ability and Lower Extremity Function, Proprioception, Trunk Control, And Balance Iduals With Stroke
Brief Title: Backward Walking and Related Factors in Individuals With Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zekiye İpek, Assoc. Prof, Gaziantep Islam Science and Technology University
Other Study IDs: ipekkirmaci..
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: stroke; back ward walking; proprioception; trunk control; balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke: Stroke Patients
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — assessment

SUMMARY:
Objective: To examine the relationship between backward walking ability and lower extremity function, proprioception, trunk control, and balance in individuals with stroke. Thirty individuals aged 30-85 who have had a stroke will be included in our study. Individuals with stroke who can walk 10 m without physical assistance, whose lower extremity functions are in the Brunnstrom motor recovery stages 2-6, who have been post-stroke for at least 3 days and up to 24 months, and who score 24 or higher on the Mini Mental Test will be included. Demographic information of individuals with stroke who meet the inclusion criteria will be recorded in a personal information form. Lower extremity function will be evaluated with the 3-meter back walking test (3MGYT), proprioception with the Fugl Meyer lower extremity assessment scale, with a digital goniometer, trunk control with the Trunk Impairment scale, and balance with the Brief BESTTest.

DETAILED DESCRIPTION:
Stroke survivors often experience lower walking performance and muscle strength than healthy individuals. Despite advances in acute stroke treatment, patients continue to require rehabilitation due to spasticity, upper and lower extremity dysfunction, shoulder and back pain, dysphagia, and deficits in mobility and gait, vision, perception, and communication. Approximately 40% of patients experience functional impairment after stroke onset, and 15-30% experience severe motor, sensory, and cognitive impairments. While some patients lose ambulation completely after stroke, in others, impaired balance reactions and increased postural sway contribute to fear of falling and an increased risk of falling. Walking backwards is necessary to perform activities of daily living, such as leaning back in a chair and opening a door. This movement can be particularly challenging for the elderly and individuals with neurological deficits. Mechanical measurements of backward walking, particularly speed, stride length, and double support base, have been noted to significantly decrease in older adults. It suggests that the inability to take effective backward steps may predispose older adults to a decrease in functional walking ability and an increased risk of falls. Therefore, we believe that identifying the factors that influence backward walking ability in stroke survivors will contribute to rehabilitation programs that include walking training. This study is the first to examine the factors that influence backward walking ability in stroke patients in relation to proprioception, trunk control, lower extremity function, and balance.

ELIGIBILITY:
Inclusion Criteria:

* who can walk 10 meters without physical assistance,
* Lower extremity functions are in stages 2-6 of the Brunnstrom motor recovery scale,
* Have been at least 3 days and no more than 24 months post-stroke,
* Scored 24 or higher on the Mini Mental Test

Exclusion Criteria:

* Individuals with neurological or orthopedic problems other than stroke that affect walking,
* A history of cardiovascular or rheumatological diseases that interfere with daily activities,
* A lower extremity lesion or fracture,
* Lower extremity spasticity of 4 on the Modified Ashworth Scale (MAS),
* Aphasia or communication disorders

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
3 meter backward walking | At baseline
  In the 3MBT, a three-meter distance will be measured on a flat surface and the start and end will be marked. The patient will be asked to walk backward when prompted to start, and will be asked to stop when prompted to stop. Individuals will be allowed to look back if they wish. For safety reasons, the tester will be allowed to walk with the patients. Measurements will be repeated three times and averaged.
Fugl-Meyer Lower Extremity Scale | At baseline
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based measure. Measurements are taken with the patient seated on a flat bed, such as a stretcher. Each parameter is scored as 0: Failure, 1: Partially Successful, and 2: Completely Successful. Motor function and sensory sections of the scale are used. The motor function assessment section is scored as 100 points, with 66 for the upper extremities and 34 for the lower extremities, and the sensory assessment section, which includes light touch and position sense, is scored as 24 points. A higher score indicates a better condition. It is a widely used, reliable, and valid test for assessing paretic upper and lower extremity motor impairments in stroke patients.
Proprioception | At baseline
  The patients' range of motion of the hip, knee, and ankle joints on the affected side is measured by fixing a digital goniometer to the joint. Data will be recorded in degrees. Patients will then be asked to half-jointly move their hip, knee, and ankle joints, without being able to see them. The difference between half of the normal joint movement and half of the joint movement performed with eyes closed will be noted. Assessments will be performed in both the prone and supine positions.
Trunk Impairment Scale | At baseline
  The Trunk Impairment Scale is a 17-item scale with three subsections that assess static sitting balance, dynamic sitting balance, and coordination. The starting position for the scale is with the individual in a 90º flexed knee, soles of the feet touching the floor, hands on the thighs, and no back support. Measurements will be repeated three times, and the individual's best results will be recorded. The lowest possible score is 0, and the highest is 23. A high score indicates good trunk control.
Brief-Bestest | At baseline
  It's a low-cost test that can be completed quickly with minimal equipment. It consists of six balance parameters. Measurements are made with a stopwatch on a flat surface. These include biomechanical constraints, stability limitations, transitions-preparatory postural alignment, reactive postural response, sensory orientation, and gait balance. Each question can be scored from a minimum of 0 to a maximum of 3, and the test can achieve a maximum of 24 points.